CLINICAL TRIAL: NCT06837064
Title: Evaluation of the Efficacy of Chatbot-based Automated Support System for Patients with Irritable Bowel Syndrome (IBS)
Brief Title: Efficacy of Chatbot for Irritable Bowel Syndrome (IBS) Patients
Acronym: IrBiS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department (Other)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Anton V. Vladzymyrskyy, Deputy Director for Research, Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-1
Record Dates: First submitted 2025-02-10; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Irritable Bowel Syndrome; Irritable Bowel Syndrome - Constipation; Irritable Bowel Syndrome - Diarrhoea; Irritable Bowel Syndrome - Mixed
Keywords: IBS; Irritable Bowel Syndrome; chatbot; eHealth
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chatbot group (Experimental): The group will receive access to the automated chatbot supporting system. Each patient will receive a unique access code (token) to register for the chatbot. Only patients with tokens present in the authorized database will be able to register, thus ensuring that the chatbot is exclusively used by study participants.
  Interventions: Device: Chatbot supporting system
- Standart care group (No Intervention): The group will receive standart care.

INTERVENTIONS:
Device: Chatbot supporting system — The intervention tool is the automated chatbot supporting system, which contains:
  A) educational information (therapeutic education and psychoeducation); B) symptom monitoring (stool quality and frequency, assessment of mood, sleep quality, physical activity, and dietary adherence on a scale of 0 to 10); C) behavioral distraction techniques, and body tension reduction techniques.
  Arms: Chatbot group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of an automated chatbot system in improving quality of life, reducing depression and anxiety, and decreasing visceral sensitivity in patients with Irritable Bowel Syndrome. The main research question is:

Is an automated chatbot as effective for patients with IBS as standard care? Participants will be asked to complete online surveys to assess quality of life, symptoms of depression and anxiety, and visceral sensitivity before and after the intervention.

DETAILED DESCRIPTION:
The study consists of three stages:

Stage 1: Patients with Irritable Bowel Syndrome (IBS) who meet the eligibility criteria will be invited to participate in the study. After providing written informed consent, all participants will be asked to complete a set of questionnaires to assess various parameters:

1. Irritable Bowel Syndrome Quality of Life (IBS-QOL);
2. Quality of Life - Short Form-36 (SF-36);
3. Symptoms of Anxiety and/or Depression - Hospital Anxiety and Depression Scale (HADS);
4. State and Trait Anxiety Levels - State-Trait Anxiety Inventory (STAI);
5. Visceral Sensitivity - Visceral Sensitivity Index (VSI);

Stage 2: Participants will be randomized into one of two groups: a chatbot group (intervention) and a standard care group (control). Prior to enrollment, both groups will receive a consultation with a gastroenterologist providing information on lifestyle, diet, and treatment. The intervention group will receive the access to a chatbot.

At the fourth and eighth week of follow-up participants in both groups will be asked to re-complete the set of questionnaires (IBS-QOL, SF-36, HADS, STAI, VSI). No routine gastroenterologist consultations will be scheduled during the follow-up period.

Stage 3: Results from the questionnaires will be analyzed and used to formulate conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years;
* Diagnosed with IBS;
* Signed informed consent.

Exclusion Criteria:

* Age under 18 years;
* Pregnant individuals;
* Patients with cognitive or sensory impairments that hinder understanding of questions in surveys, scales, or instruments used in the study;
* Patients unable to use a chatbot;
* Patients currently participating in any other clinical trial or experimental study;
* Patients with psychotic symptoms;
* Patients with other conditions that may influence the endpoints of the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change the Health-related quality of life in IBS | 8 weeks
  Change the quality of life in IBS according to Irritable Bowel Syndrome Quality of Life (IBS-QOL) questionnaire. The IBS-QOL is a self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment. Max score is 100, min score is 0.
  Higher score means better outcome
Change the Health-related quality of life in IBS | 8 weeks
  Change the quality of life in IBS according to Short Form-36 (SF-36) questionnaire. The questionnaire consists of 8 sections:
  * Vitality;
  * Physical functioning;
  * Bodily pain;
  * General health perceptions;
  * Physical role functioning;
  * Emotional role functioning;
  * Social role functioning;
  * Mental health; For each section scores range from 0 to 100. Lower scores mean more disability, higher scores mean less disability.

SECONDARY OUTCOMES:
Change psychological well-being of patients with IBS measured by HADS | 8 weeks
  Change psychological well-being of patients with IBS according to Hospital Anxiety and Depression Scale (HADS). Each item is scored on a response-scale with four alternatives ranging between 0 and 3. Score 8-10 for doubtful cases and ≥11 for definite cases of depression and anxiety.
Change psychological well-being of patients with IBD measured by VSI | 8 weeks
  Change psychological well-being of patients with IBD according to Visceral Sensitivity Index (VSI). Min value is 0, max value is 75. 0-10 - no GI-specific anxiety; 11-30 - moderate GI-specific anxiety; 31 - 75 - severe GI-specific anxiety; Lower score means better outcome.
Change psychological well-being of patients with IBS measured by STAI | 8 weeks
  Change psychological well-being of patients with IBS measured by State-Trait Anxiety Inventory (STAI) questionnaire. The STAI has 20 items to assess trait anxiety and 20 to assess state anxiety. The score range for each subscale is 20-80, the higher score indicating anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Anton V. Vladzymyrskyy, PhD, Study Director — Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department
Locations (1):
- Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided